CLINICAL TRIAL: NCT01539265
Title: A Randomized, Double-blind, Placebo-controlled, Phase II Study of Silodosin in Patients With Urinary Calculi
Brief Title: A Dose-finding Study of Silodosin in Patients With Urinary Calculi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMD3201
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Calculus
Keywords: urinary calculus; ureteral stones; medical expulsive therapy
MeSH Terms: conditions — Urinary Calculi | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- silodosin, arm 1 (Experimental)
  Interventions: Drug: silodosin
- silodosin, arm 2 (Experimental)
  Interventions: Drug: silodosin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: silodosin
  Arms: silodosin, arm 1
Drug: silodosin
  Arms: silodosin, arm 2
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of silodosin in urinary calculi patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a unilateral ureteral calculus with ≥ 5 mm and ≤ 10 mm at Week 0.
* Patients who are able to visit the site continually as out-patient during the study

Exclusion Criteria:

* Patients who have multiple urethral stones.
* Patients who have or have history of a ureteral stricture or other structural passage obstruction of the ureter on affected side.
* Patients who have been diagnosed with myasthenia gravis, myopathy, spina bifida, spinal cord injury, or fibromyalgia syndrome.
* Patients who have a clinically significant hepatic or renal disorder.
* Patients with postural hypotension or with a history of postural hypotension.
* Patients with a history of sever drug allergy, or patients with a history of hypersensitivity to silodosin.
* Patients who are pregnant, nursing, or desire pregnancy during the study period, or patients who cannot strictly comply with a physician's contraception directions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

PRIMARY OUTCOMES:
Spontaneous stone passage rate | 4 weeks

SECONDARY OUTCOMES:
Time to spontaneous stone passage | 4 weeks
Analgesic use | 4 weeks
Pain severity | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Clinical Development Department, Kissei pharmaceutical Co., Ltd.
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan